CLINICAL TRIAL: NCT06273696
Title: Evaluation of the Acceptability and Safety of the ShangRing Device for Male Circumcision in Shinyanga, Tanzania
Status: Completed | Type: Observational
Sponsor: IntraHealth International (Other)
Collaborators: Ministry of Health, Tanzania (Other Government); President Office Regional Administration and Local Government, Tanzania (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Jhpiego (Other); World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-519; NU2GGH001927 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2023-02-09; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Penile Infection; Penile Haematoma; Penile Bleeding; Deformity
Keywords: male circumcision; ShangRing; adverse events; Tanzania; HIV/AIDS; nonsurgical circumcision; voluntary medical male circumcision; device; anesthesia
MeSH Terms: conditions — Congenital Abnormalities; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 49 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Circumcision clients: Participants who underwent the ShangRing circumcision procedure
  Interventions: Device: ShangRing

INTERVENTIONS:
Device: ShangRing — The ShangRing is a sterile, single use, disposable male circumcision (MC) device that consists of two concentric plastic rings, the inner of which is lined by a silicone pad, which provides a smooth and non-bio reactive surface against the surgical wound. The outer ring consists of 2 halves which are hinged together at the same end. On each side of the halves there is a locking clasp which allows for locking itself with inner ring. The ShangRing device is removed seven days after placement.

SUMMARY:
The goal of this observational study was to evaluate the safety and acceptability of the ShangRing device for male circumcision among men in Shinyanga, Tanzania. The main question aims to answer both provider acceptability (practicality of device use and placement and removal times) and client acceptability (comfort during placement and removal, experience while wearing the ring, and penile appearance after healing). Participants voluntarily underwent male circumcision using the ShangRing device and before being discharged, were interviewed about their experience. Participants were also interviewed at device removal day (day 7), during a follow-up phone call (day 10), a sample were selected to participate in in-depth interviews (day28), and finally all men were asked to return for a follow-up visit (day 49).

DETAILED DESCRIPTION:
Medical circumcision devices have the potential to accelerate delivery of male circumcision by making the procedure quicker and easier, while remaining as safe as surgical circumcision. Thus, circumcision devices may facilitate expansion of adult male circumcision programs for HIV prevention and address some of the common capacity issues in the U.S. President's Emergency Plan for AIDS Relief (PEPFAR) priority countries for male circumcision.

One promising device for adult male circumcision is ShangRing, which was prequalified by the World Health Organization (WHO) in 2015 for males aged 13 and older. WHO has created a framework for introducing circumcision devices in a country. This framework recommends countries take a methodical approach to introducing circumcision devices, evaluating acceptability and safety within its health system before making widespread adoption.

Evaluation Goal: To evaluate the safety and acceptability of the ShangRing device for nonsurgical circumcision in routine clinical settings, as a part of a comprehensive HIV prevention program for males in voluntary medical male circumcisions (VMMC) programs.

Evaluation Endpoints: the proportion of males experiencing mild, moderate and severe adverse events (AEs) associated with ShangRing circumcision procedures, including both intra- and post-operative events, and all device-related malfunctions (e.g., early spontaneous detachment).

Evaluation Design

Training Phase: this phase was used to evaluate the training requirements for implementation by mid-level providers, to preliminarily assess acceptability to providers, and to monitor logistical needs. Each clinician performed no fewer than 10 ShangRing device placements, and 5 ShangRing removals before start of the next phase (implementation pilot).

Implementation Pilot: following the training period, 575 male clients were recruited to undergo circumcision with the ShangRing device in the context of routine service delivery.

Data was collected at up to at least 5 points in time: at enrollment and device placement (day 0), at device removal (day 7), during a follow-up phone call (day 10), in-depth qualitative interviews for 50 purposefully selected clients (day 28), at an in-person follow-up visit to assess wound healing (day 49), and at subsequent weekly visits to assess healing for those not completely healed at day 49. Upon completion of the implementation pilot, the data was analyzed and used to assist with policy decisions and recommendations on ShangRing use in adult male circumcision programs.

ELIGIBILITY:
Inclusion Criteria:

* Be an uncircumcised male aged 13 years or older
* Be seeking medical circumcision at one of the study sites
* Consent to an HIV test, unless they were known to be HIV-positive
* Agree to be circumcised using the ShangRing device
* Have their penis fit into one of the ShangRing ring sizes available during the study
* Be able to understand the evaluation procedures and requirements
* Agree to abstain from sexual intercourse and masturbation for six weeks after ring removal, for a total of seven weeks
* Live within 30 kilometers of the facility in Shinyanga Region, Tanzania
* Be willing to provide valid contact information (i.e., telephone number, address of residence, place of employment, and other locator information) and be willing to receive communications and/or follow-up visits
* Have an activated mobile phone or access to a mobile phone
* Agree to return for a follow-up visit to assess healing at day 49 (42 days post-removal)
* Agree to a ten-day post-placement (three days post-removal) telephone call to assess and detect symptoms of AEs
* Be able to communicate in English and/or Kiswahili
* Be capable and willing to provide written informed consent (18 years and older) or written informed consent from a parent guardian (13-17 years) to participate for both HIV testing services and VMMC services

Exclusion Criteria:

* A cognitive impairment that prevented the client from providing consent
* Any health condition (reported or observed) that was a contraindication to surgical VMMC in the national program or that ShangRing providers deemed a contraindication.

These may include diabetes, peripheral vascular disease, cancer, bleeding disorders, and/or current moderate or severe infectious illness.

* A current sexually transmitted infection (STI) other than HIV (clients with STIs were advised to return for circumcision once the STI was treated); and/or other conditions, which in the opinion of the site supervisor, prevented the client from undergoing a circumcision with the ShangRing device.

Min Age: 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Men and boys who choose to undergo voluntary medical male circumcision
Study Population: Shinyanga is one of the 31 regions, in the Lake Zone Region of Tanzania. Shinyanga covers a total of 18,555 square kilometers. As of the 2012 census, the population of the Shinyanga region was 1,534,808. The economy of the region is primarily driven by agriculture. As of 2011, the HIV prevalence of Shinyanga was 7.4%. According to the Tanzania Demographic Health Survey and Malaria Indicator Survey, 54% of men in Shinyanga reported that they are circumcised.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 49 days post device placement
  Total numbers and types of known adverse events (AE)s occurring among clients, including all severities of AEs (mild, moderate, severe) and serious AEs, including detailed information about all instances of device displacement/detachment/self-removal/malfunction, need for medical attention or intervention, and final outcomes in those experiencing AEs
Number of Clients with Adverse Events | 49 days post device placement
  Total number of clients with known adverse events (AEs) (may be different from above if clients experience multiple AEs), including all severities of AEs and serious AEs
Descriptions of Adverse Events | 49 days post device placement
  A description of each adverse event by type and classification, severity, time of occurrence (during placement, in situ, or during removal) time of detection (days post-application and/or post-removal) captured as date AE is diagnosed, clinical management, and resolution

SECONDARY OUTCOMES:
Provider Training | 49 days post device placement
  Determine the training needed for proficiency, including number of procedures required under supervision to become certified as fully proficient. This will involve analyzing AE rates stratified by during training and post-training in addition to overall.
Client Follow-up Visit Rate | 49 days post device placement
  Total number of clients who return for recommended follow-up at 49 days post-device placement, divided by the total number of ShangRing-circumcised clients
Client Preference for ShangRing Over Surgical Circumcision | At device removal (7 days post device placement)
  Proportion of ShangRing clients who report they would still choose ShangRing method over surgical circumcision. This was captured using multiple choice:
  "After having worn the ring for a week, would you still choose ShangRing for circumcision, or would you choose surgery?"
  1. I would definitely choose ShangRing again
  2. I would probably choose ShangRing again
  3. I would probably choose surgery
  4. I would definitely choose surgery
  5. I don't know
Client Recommendation Rate | At device removal (7 days post device placement)
  Proportion of clients who report they would recommend VMMC using ShangRing. This was captured with a yes/no question:
  "At this point would you recommend ShangRing to someone you know who is considering circumcision?" Yes No I don't know
Cosmetic Result Acceptability | At device removal (7 days post device placement)
  Client reporting on the cosmetic result post-removal. This was captured with multiple choice:
  "How satisfied are you with the appearance of your penis?"
  1. I am very satisfied
  2. I am satisfied
  3. I am dissatisfied
  4. I am very dissatisfied
  5. I don't know
Client Experience While Performing Routine Activities | At device removal (7 days post device placement)
  Client reports on their experience while wearing ShangRing. This is captured with multiple choice:
  "How much did the ring affect you while performing day-to-day activities?"
  1. It did not affect me at all
  2. It only affected me while performing certain activities
  3. It affected me during all activities, but I could still do them
  4. It prevented me from performing certain activities
Client Discomfort | At device removal (7 days post device placement)
  Clients' opinions discomfort while wearing the ShangRing. This was captured with multiple choice:
  "How much discomfort did you experience while wearing the ShangRing device over the past seven days?"
  1. I had no discomfort while wearing the ring
  2. I had minor discomfort while wearing the ring
  3. I had moderate discomfort while wearing the ring
  4. I had a lot of discomfort while wearing the ring
Provider Ease of Application | Immediately after the completion of the provider ShangRing training
  Provider perceived ease of application, captured with a Likert scale:
  "I found ShangRing circumcisions to be easy to perform."
  1. Strongly disagree
  2. Disagree
  3. Neither Agree nor Disagree
  4. Agree
  5. Strongly Agree
Provider Preference | Immediately after the completion of the provider ShangRing training
  Provider perceived preference of performing ShangRing procedures, captured with a Likert scale:
  "I prefer performing ShangRing procedures over surgical circumcision."
  1. Strongly disagree
  2. Disagree
  3. Neither Agree nor Disagree
  4. Agree
  5. Strongly Agree
Provider Recommendation | Immediately after the completion of the provider ShangRing training
  Provider recommendation of ShangRing to potential clients, captured with a Likert scale:
  "I would advise that clients select ShangRing circumcision over surgical circumcision."
  1. Strongly disagree
  2. Disagree
  3. Neither Agree nor Disagree
  4. Agree
  5. Strongly Agree
Description of Procedures | 49 days post device placement
  Measure both the ShangRing application and removal times, including the time it took for topical anesthesia to take effect
Healing rate | 52 days post device placement
  The percentage of clients determined by a clinician to be clinically healed 49-52 days post-placement of the ShangRing device (42 days post-removal), and the time at which point all clients are clinically healed

CONTACTS AND LOCATIONS:
Overall Officials: Lija Gissenge, MD, MMed, Principal Investigator — Head, HIV Prevention Unit, Tanzania Ministry of Health, Community Development, Gender and Children
Locations (2):
- Tanzania (2):
  - Kahama District Hospital, Shinyanga
  - Ushetu Health Centre, Shinyanga

IPD SHARING:
Plan to Share IPD: No
Per our data sharing agreement with the Tanzania Ministry of Health (MOH) and the local institutional review board (IRB) Ethics Review Committee, we are not authorized to share individual patient information with anyone outside the study team.

REFERENCES:
- [Background] Auvert B, Taljaard D, Lagarde E, Sobngwi-Tambekou J, Sitta R, Puren A. Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial. PLoS Med. 2005 Nov;2(11):e298. doi: 10.1371/journal.pmed.0020298. Epub 2005 Oct 25. PMID 16231970
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Bailey RC, Moses S, Parker CB, Agot K, Maclean I, Krieger JN, Williams CF, Campbell RT, Ndinya-Achola JO. Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial. Lancet. 2007 Feb 24;369(9562):643-56. doi: 10.1016/S0140-6736(07)60312-2. PMID 17321310
- [Background] WHO Prequalification of Male Circumcision Devices Public Report. Product: ShangRing. WHO reference number: PQMC 0003-003-00. March 2019, version 3.0.
- [Background] Peng YF, Cheng Y, Wang GY, Wang SQ, Jia C, Yang BH, Zhu R, Jian SC, Li QW, Geng DW. Clinical application of a new device for minimally invasive circumcision. Asian J Androl. 2008 May;10(3):447-54. doi: 10.1111/j.1745-7262.2008.00411.x. PMID 18385906
- [Background] Cheng Y, Peng YF, Liu YD, Tian L, Lu NQ, Su XJ, Yan ZJ, Hu JS, Lee R, Kim HH, Sokal DC, Li PS. [A recommendable standard protocol of adult male circumcision with the Chinese Shang Ring: outcomes of 328 cases in China]. Zhonghua Nan Ke Xue. 2009 Jul;15(7):584-92. Chinese. PMID 19694369
- [Background] Barone MA, Li PS, Awori QD, Lee R, Goldstein M. Clinical trials using the Shang Ring device for male circumcision in Africa: a review. Transl Androl Urol. 2014 Mar;3(1):113-24. doi: 10.3978/j.issn.2223-4683.2014.01.09. PMID 26816759
- [Background] Barone MA, Awori QD, Li PS, Simba RO, Weaver MA, Okech JO, Aduda AO, Cherutich P, Muraguri N, Wekesa JM, Nyanchoka J, Perchal P, Masson P, Lee R, Goldstein M, Kioko J, Lusi O, Sokal DC. Randomized trial of the Shang Ring for adult male circumcision with removal at one to three weeks: delayed removal leads to detachment. J Acquir Immune Defic Syndr. 2012 Jul 1;60(3):e82-9. doi: 10.1097/QAI.0b013e31824ea1f2. PMID 22343180
- [Background] Sokal DC, Li PS, Zulu R, Awori QD, Combes SL, Simba RO, Lee R, Hart C, Perchal P, Hawry HJ, Bowa K, Goldstein M, Barone MA. Randomized controlled trial of the shang ring versus conventional surgical techniques for adult male circumcision: safety and acceptability. J Acquir Immune Defic Syndr. 2014 Apr 1;65(4):447-55. doi: 10.1097/QAI.0000000000000061. PMID 24583615
- [Background] Barone MA LP, Zulu R, Awori QD, et al. A Field Study of Male Circumcision Using the Shang Ring, a Minimally Invasive Disposable Device, in Routine Clinical Settings in Kenya and Zambia. 7th International AIDS Society Conference on HIV Pathogenesis, Treatment and Prevention; Kuala Lumpur, Malaysia, 2013.
- [Background] Kigozi G, Musoke R, Watya S, Kighoma N, Ssebbowa P, Serwadda D, Nalugoda F, Makumbi F, Li P, Lee R, Goldstein M, Wawer M, Sewankambo N, Gray RH. The acceptability and safety of the Shang Ring for adult male circumcision in Rakai, Uganda. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):617-21. doi: 10.1097/QAI.0b013e3182968dda. PMID 23614991
- [Background] Rech D, Bertrand JT, Thomas N, Farrell M, Reed J, Frade S, Samkange C, Obiero W, Agot K, Mahler H, Castor D, Njeuhmeli E. Surgical efficiencies and quality in the performance of voluntary medical male circumcision (VMMC) procedures in Kenya, South Africa, Tanzania, and Zimbabwe. PLoS One. 2014 May 6;9(5):e84271. doi: 10.1371/journal.pone.0084271. eCollection 2014. PMID 24802412
- [Background] Bratt JH, Zyambo Z. Comparing direct costs of facility-based Shang Ring provision versus a standard surgical technique for voluntary medical male circumcision in Zambia. J Acquir Immune Defic Syndr. 2013 Jul 1;63(3):e109-12. doi: 10.1097/QAI.0b013e31828e9526. PMID 23481667
- [Background] Sokal DC, Li PS, Zulu R, Awori QD, Agot K, Simba RO, Combes S, Lee RK, Hart C, Lai JJ, Zyambo Z, Goldstein M, Feldblum PJ, Barone MA. Field study of adult male circumcision using the ShangRing in routine clinical settings in Kenya and Zambia. J Acquir Immune Defic Syndr. 2014 Dec 1;67(4):430-7. doi: 10.1097/QAI.0000000000000321. PMID 25162816
- [Background] Tanzania Commission for AIDS (TACAIDS), Zanzibar AIDS Commission (ZAC). Tanzania HIV Impact Survey (THIS) 2016-2017: Final Report. Dar es Salaam, Tanzania. December 2018.
- [Background] The United Republic of Tanzania, Voluntary medical male circumcision country operational plan: 2014-2017. November 2014.
- [Background] Preventing HIV Through Safe Voluntary Medical Male Circumcision for Adolescent Boys and Men in Generalized HIV Epidemics: Recommendations and Key Considerations. Geneva: World Health Organization; 2020 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK562463/ PMID 32986340
- [Background] Kigozi G, Musoke R, Kighoma NGR. The acceptability and safety of the ShangRing for adolescent male circumcision in Rakai, Uganda. International AIDS Society Conference; 2014; Melbourne, Australia. TUPE148 p.
- [Background] Awori QD, Lee RK, Li PS, Moguche JN, Ouma D, Sambai B, Goldstein M, Barone MA. Use of the ShangRing circumcision device in boys below 18 years old in Kenya: results from a pilot study. J Int AIDS Soc. 2017 Jul 12;20(1):21588. doi: 10.7448/IAS.20.1.21588. PMID 28715157
- See also: The Joint United Nations Programme on HIV/AIDS (UNAIDS). Fast track commitments to end AIDS by 2030. — http://www.unaids.org/sites/default/files/media_asset/fast-track-commitments_en.pdf
- See also: Tetanus and VMMC: risk according to circumcision method and risk mitigation. Report of the WHO Technical Advisory Group on Innovations in Male Circumcision - consultative review of additional information, 12 August 2016. — https://www.who.int/publications/i/item/WHO-HIV-2016.19
- See also: Project Improving Quality VMMC (IQ) Virtual Seminar series. Virtual Roundtable on ShangRing for VMMC: Country perspectives. September 9th 2019. — http://www.malecircumcision.org/resource/introduction-virtual-roundtable-shangring-vmmc-country-perspectives
- See also: PEPFAR Dashboards. Country and Regional Program Results, Fiscal Year (FY) 2010-2016: Tanzania. May 5, 2017. — http://data.pepfar.net/country/impact?country=Tanzania&indicatorGroup=HIV%20Prevention&year=2004&yearTo=2016.
- See also: World Health Organization. Framework for clinical evaluation of devices for male circumcision. September 2012. — http://apps.who.int/iris/bitstream/10665/75954/1/9789241504355_eng.pdf?ua=1
- See also: World Health Organization. Manual for male circumcision under local anesthesia and HIV prevention services for adolescent boys and men (2018). — https://www.who.int/publications/i/item/manual-for-male-circumcision-under-local-anaesthesia-and-hiv-prevention-services-for-adolescent-boys-and-men

DOCUMENTS (2):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT06273696/Prot_000.pdf
  • Informed Consent Form (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT06273696/ICF_001.pdf